CLINICAL TRIAL: NCT02585856
Title: Efficacy and Safety of Photodynamic Therapy for Unresectable Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, associate director, First People's Hospital of Hangzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-001-02
Record Dates: First submitted 2015-10-01; First posted 2015-10-23 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cholangiocarcinoma
Keywords: Biliary duct carcinoma; Photodynamic therapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDT+stent (Experimental): Patients with unresectable CCA are performed PDT and biliary stent with ERCP
  Interventions: Device: PDT; Device: stent
- stent (Placebo Comparator): Patients with unresectable CCA are performed biliary stent with ERCP alone
  Interventions: Device: stent

INTERVENTIONS:
Device: PDT — Patients with unresectable CCA are performed PDT with ERCP after porfimer sodium （chongqing ray high medical instrument co., LTD，Chongqing, China) i.v. at a dose of 2 mg/kg at 48 h.
  PDT procedure: for light distribution, flexible cylindrical diffuser probes mounted on 400-mm quartz fibres with an active distal tip length of 2 cm （chongqing ray high medical instrument co., LTD，Chongqing, China) is used. The light source was a diode laser system with a maximum power output of 2 Wand a wavelength of 633.3 nm. The power emitted by the diffuser tip was calibrated to 400 mW/cm before PDT was administered using an integrating sphere power meter. The mean irradiation time was 452 s (range: 400-600 s), using a power density of 300-400 mW/cm and an energy dose of 180-200 J/cm (of diffuser length).
  Arms: PDT+stent
Device: stent — Patients with unresectable CCA are performed with ERCP, one or several plastic biliary stents (Boston Scientific Corporation, MA,USA) are inserted to ensure adequate decompression and bile drainage.

SUMMARY:
The aim of this study is to investigate the efficacy of photodynamic therapy (PDT) in increasing the survival time, decreasing cholestasis and improving health-related quality of life (HRQoL) by comparing PDT puls stents versus stents alone in patients with unresectable cholangiocarcinoma,and to assess the safety of PDT by observing the complications after the procedure.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is difficult to diagnose due to its anatomic location, clinical course, and lack of definitive diagnostic criteria. It is often clinically silent with symptoms developing only in advanced disease. Surgical resection is the recommended curative intervention with only a minority of patients (10-20%) having potentially resectable tumors at time of diagnosis.

Endoscopic palliative therapy in CCA entails the relief of obstructive jaundice through transpapillary or percutaneous insertion of plastic or metal biliary stents. Although biliary decompression provides relief of cholangitis and improvement in quality of life, it does not improve survival.

Photodynamic therapy (PDT) in conjunction with biliary stenting may improve bile duct patency by local obliteration of malignant tissue through the cytotoxic effects of reactive oxygen species. Several studies suggest PDT plus biliary stent placement may prolong survival (range of 360-630 days), reduce cholangitis, and improve the quality of life of patients with advanced disease. The aim of this study is to determine the effectiveness and safety of PDT with biliary stenting compared to biliary stenting alone in the palliative treatment of unresectable CCA in China.

ELIGIBILITY:
Inclusion Criteria:

* Obtention of a written informed consent.
* Patient over 18.
* Patient with histologically proved cholangiocarcinoma ; histologic diagnosis must be proved by biliary brushing, bile cytology, endobiliary biopsy under Spyglass, or by EUS-FNA.
* Patient with Karnofsky score ≥ 50 %
* Patient capable of fill in the quality of life questionnaire

Exclusion Criteria:

* No written informed consent.
* Patients under or already treated by radiotherapy or chemotherapy treatment for cholangiocarcinoma.
* Patients with porphyria or hypersensibility to porphyrins.
* Pregnant, parturient or breastfeeding women.
* Patient under 18.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-02; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
survival time | two years

SECONDARY OUTCOMES:
clinical success rates | two years
  The proportion of patients whose bilirubin decreased obviously after procedure
Karnosky performance status score | two years
complications | two years
  Number of patients with complications,type, frequency and intensity of complications between this two group will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.S, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
publication

REFERENCES:
- [Background] Rustagi T, Jamidar PA. Endoscopic treatment of malignant biliary strictures. Curr Gastroenterol Rep. 2015 Jan;17(1):426. doi: 10.1007/s11894-014-0426-9. PMID 25613178
- [Result] Wagner A, Kiesslich T, Neureiter D, Friesenbichler P, Puespoek A, Denzer UW, Wolkersdorfer GW, Emmanuel K, Lohse AW, Berr F. Photodynamic therapy for hilar bile duct cancer: clinical evidence for improved tumoricidal tissue penetration by temoporfin. Photochem Photobiol Sci. 2013 Jun;12(6):1065-73. doi: 10.1039/c3pp25425a. Epub 2013 Apr 4. PMID 23558738
- [Result] Lee TY, Cheon YK, Shim CS, Cho YD. Photodynamic therapy prolongs metal stent patency in patients with unresectable hilar cholangiocarcinoma. World J Gastroenterol. 2012 Oct 21;18(39):5589-94. doi: 10.3748/wjg.v18.i39.5589. PMID 23112552
- [Result] Kahaleh M. Photodynamic therapy in cholangiocarcinoma. J Natl Compr Canc Netw. 2012 Oct 1;10 Suppl 2:S44-7. doi: 10.6004/jnccn.2012.0174. PMID 23055215
- [Result] Leggett CL, Gorospe EC, Murad MH, Montori VM, Baron TH, Wang KK. Photodynamic therapy for unresectable cholangiocarcinoma: a comparative effectiveness systematic review and meta-analyses. Photodiagnosis Photodyn Ther. 2012 Sep;9(3):189-95. doi: 10.1016/j.pdpdt.2012.03.002. Epub 2012 Apr 11. PMID 22959798